### The GlaxoSmithKline group of companies

| Division | | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : Phase I, single-center, open label, fixed-sequence cross-<br>study to evaluate the effect of rifabutin on the<br>pharmacokinetics of oral cabotegravir in healthy subject | |
|---|---|---|
| <b>Compound Number</b> | : | GSK1265744 |
| <b>Effective Date</b> | : | 08-SEP-2017 |

## **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Pharmacology Study Report for Protocol 205712
- This RAP is intended to describe the safety, pharmacokinetics (PK), and tolerability analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

### RAP Author(s):

| Approver | Date | Approval<br>Method |
|---|---|---|
| Associate Director, Clinical Statistics, PAREXEL | 07-SEP-2017 | email |
| Director, Clinical Pharmacology Modelling & Simulation, GSK | 08-SEP-2017 | email |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## The GlaxoSmithKline group of companies

## **RAP Team Approvals:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| PPD | 30-AUG-2017 | email |
| Clinical Program Lead, PCPS CPSSO, GSK | | |
| PPD | 31-AUG-2017 | email |
| Director, Clinical Development, ViiV Physicians | | |
| PPD | 05-SEP-2017 | email |
| Principal Data Manager (CPSSO Data<br>Management GSK) | | |
| PPD | | email |
| Principal Statistical Programmer (Statistical programming, PAREXEL) | 07-SEP-2017 | |
| Director, (ViiV, Clinical Pharmacology) | 30-AUG-2017 | email |

## **Clinical Statistics and Clinical Programming Line Approvals:**

| Approver | Date | Approval<br>Method |
|---|---|---|
| Manager, Statistics (Infection Disease, Clinical Statistics GSK) | 31-AUG-2017 | email |
| Programming Manager, (ID, Clinical Programming, GSK) | 31-AUG-2017 | email |

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | INTRO | DUCTIO | N | 5 |
| 2. | SUMM | IARY OF | KEY PROTOCOL INFORMATION | 6 |
| | 2.1. | | to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | Study Ok | pjective(s) and Endpoint(s) | 6 |
| | 2.3. | Study De | esign | <mark>7</mark> |
| | 2.4. | | al Hypotheses | |
| 3. | PLANI | | LYSIS | |
| | 3.1. | | nalyses | |
| | 3.2. | Final Ana | alyses | 8 |
| 4. | ANAL' | | PULATIONS | |
| | 4.1. | Protocol | Deviations | 9 |
| 5. | | | ONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONV | ENTIONS | S | 10 |
| 6. | STUD | Y POPUL | ATION ANALYSES | 10 |
| • | 6.1. | | v of Planned Analyses | |
| 7 | | NDV OTAT | TISTICAL ANALYSES | 44 |
| 7. | 7.1. | | cokinetic Analyses | |
| | 7.1. | 7.1.1. | Overview of Planned Pharmacokinetic Analyses | |
| | | 7.1.2. | Drug Concentration Measures | 12 |
| | | 7.1.3. | Pharmacokinetic Parameters | |
| | 7.2. | Statistica | al Analysis of Pharmacokinetic Parameters | |
| 8. | SECO | NDARY S | STATISTICAL ANALYSES | 14 |
| ٠. | 8.1. | | nalyses | |
| | | | Overview of Planned Analyses | |
| 9. | REFE | RENCES. | | 16 |
| 40 | | NDIOEO | | 47 |
| 10. | | | x 1: Protocol Deviation Management | |
| | 10.1. | 10 1 1 | Exclusions from PK Parameter Summary Population | 10<br>10 |
| | 10.2. | Annendi | x 2: Data Management | 10 |
| | 10.2. | 10.2.1. | —————————————————————————————————————— | |
| | 10.3. | - | x 3: Time & Events | |
| | | 10.3.1. | | |
| | 10.4. | Appendix | x 4: Treatment States and Phases | 24 |
| | | 10.4.1. | Treatment State and Study Phases | 24 |
| | | | 10.4.1.1. Treatment States for AE, SAE and | _ |
| | | | Concomitant Medications Data | |
| | 40.5 | A m.m :!' | 10.4.1.2. Reporting Other Safety Data | |
| | 10.5. | Appendix<br>10.5.1. | x 5: Data Display Standards & Handling Conventions Study Treatment & Sub-group Display Descriptors | |
| | | 10.5.1. | | |

### CONFIDENTIAL

| | | 10.5.2.1. | Baseline Definitions | .26 |
|---|---|---|---|---|
| | | 10.5.2.2. | Derivations and Handling of Missing Baseline | |
| | | | Data | . 27 |
| | 10.5.3. | Reporting | Process & Standards | . 27 |
| 10.6. | Appendix | 6: Derived | and Transformed Data | . 30 |
| | 10.6.1. | General | | . 30 |
| | 10.6.2. | • | ulation | |
| | 10.6.3. | | | |
| 10.7. | | | ure Withdrawals & Handling of Missing Data | |
| | 10.7.1. | | Withdrawals | |
| | 10.7.2. | | f Missing Data | |
| | | | Handling of Missing Dates | |
| | | | Handling of PK Concentration Data | |
| 10.8. | | | of Potential Clinical Importance | |
| | 10.8.1. | | Values | |
| | 10.8.2. | | | |
| | | | <u></u> | |
| 10.9. | • • | | Specifications for Statistical Analysis | |
| | 10.9.1. | | Analysis Assumptions and Model Specifications | |
| 10.10. | | | eviations & Trade Marks | |
| | | | ons | |
| | | | (S | |
| 10.11. | | | Data Displays | |
| | | | ay Numbering | |
| | | | mple Referencing | |
| | | , | ulation Tables | |
| | | , | oles | |
| | | | kinetic Tables | |
| | | | kinetic Figures | |
| | | | gs | |
| | | | istings | |
| 10.12. | | | ole Mock Shells for Data Displays | |
| | 10.12.1. | Data Displ | ay Numbering | .47 |

## 1. INTRODUCTION

The purpose of this reporting and analysis plan (RAP) is to describe the analyses to be included in the Clinical Study Report for Protocol 205712:

| Revision Chronology: | Revision Chronology: | |
|---|---|---|
| GSK Document No.: 2016N269788_00 | 23-FEB-2017 | Original |
| GSK Document No.:<br>2016N269788_01 | 13-APR-2017 | The purpose of this protocol amendment is to update Appendix 12.5.1." Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential(FRP)". The updates include clarifying true abstinence for this study and the deletion of double barrier method: condom and occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent foam/gel/film/cream/suppository) as a highly effective method for avoiding pregnancy in females of reproductive potential (FRP) |
| GSK Document No.:<br>2016N269788_02 | 29-JUN-2017 | Clarify the required days for fasting (Day 14 and Day 28). Remove Appendix 12.4.3- Definition of Cardiovascular Events. The collection of Cardiovascular Events is not applicable to the 205712 study. |

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

### **Changes to the Protocol Defined Statistical Analysis Plan** 2.1.

There were no changes or deviations to the originally planned statistical analysis specified in the protocol amendment 2 (Dated: 29-Jun-2017).

#### Study Objective(s) and Endpoint(s) 2.2.

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| To compare steady state CAB exposure following 30 mg oral dose once daily with and without RBT 300 mg once daily. | • Plasma CAB AUC(0-τ), Cmax |
| Secondary Objectives | Secondary Endpoints |
| To describe the pharmacokinetic (PK) of<br>CAB 30 mg oral dose once daily<br>administered alone and co-administered<br>with RBT. | • Plasma CAB Cτ, tmax, t1/2 and CL/F |
| To assess the safety and tolerability of<br>CAB 30 mg oral dose administered<br>alone and in combination with RBT<br>300 mg once daily. | Safety and tolerability parameters, including adverse events, concurrent medication, clinical laboratory screens, electrocardiogram (ECG), and vital signs assessments. |
| AUC <sub>(0-t)</sub> = area under the plasma concentration time curve from time zero to the last quantifiable time point | |

C<sub>max</sub> = maximum observed concentration

Ct = last quantifiable concentration

t<sub>max</sub> = time of maximum observed concentration

 $t_{1/2}$  = the elimination half-lifeCL/F = apparent oral clearance

# 2.3. Study Design

| ( | Overview of Study Design and Key Features | | | | |
|---|---|---|---|---|---|
| T | able 1 | Study Design | | | |
| | Subjects | Screening Period | Period 1<br>Days 1 – 14 | Period 2<br>Days 15 - 28 | Follow-up |
| | N=15 | Within 30 Days of Day 1 | Treatment A | Treatment B | ~10-14 days after<br>last dose of CAB |
| • | | A = CAB 30 mg once daily x | • | | |
| • | | B = RBT 300 mg once daily | | | 2 : 1 |
| | Design | | | , open label, fixed-se | equence, 2-period |
| | Subjects will undergo a screening visit within 30 days of the first dose of study drug, followed by two treatment periods and a follow-up period. • Approximately 15 healthy adult subjects will be enrolled to ensure that 12 subjects will complete dosing and critical assessments. • Period 1: Eligible participants will be admitted to the unit on Day -1. Subjects will be dosed for Days 1, 13 and 14 under the fasting conditions in the unit and subjects will be dispensed a bottle of CAB to be taken at home on Days 2-12 and discharged from the unit. Subjects will be provided with a subject diary to document daily recordings of dosing occurring outside of the unit. There will be no washout between Period 1 and Period 2. • Period 2: On Day 15 following the completion of the required Day 14 safety assessments and PK collection, subjects will proceed to Period | | | ow-up period. Illed to ensure essments. e unit on Day -1. he fasting a bottle of CAB on the unit. ment daily here will be no e required Day 14 roceed to Period of T 300 mg and a | |
| <ul> <li>2, where site staff will administer a single dose of RBT 300 mg and a single dose of CAB 30 mg after an overnight fast of at least 6 hours in the unit. Subjects will be discharged and dispensed a bottle of RBT and a bottle of CAB to be taken at home on Days 16-20 and 22-25. Subjects will be provided with a subject diary to document daily recordings of home dosing. In the morning of Days 21, subjects will bring their bottle of RBT and bottle of CAB for observed dosing in the unit and safety assessments as an outpatient visit. On Days 26 and 27, subjects will return to the unit for a pre-dose PK collection and observed dosing as an outpatient visit and then be discharged home. In the morning of Day 28 following an overnight fast of at least 6 hours, subjects will receive a single dose of RBT and a single dose of CAB in the unit with serial CAB PK samples collected pre-dose and through 24 hours after dosing up to Day 29.</li> <li>Subjects will be discharged from the unit on Day 29 after the final assessment is completed. Subjects will complete a follow-up visit ~ 10-14 days after the last 30 mg oral dose of CAB.</li> </ul> | | | | | |

| Overview of S | Overview of Study Design and Key Features |
|---|---|
| Treatment<br>Assignment | <ul> <li>Subjects will receive following treatments in a fixed sequence of A/B:</li> <li>Treatment A = CAB 30 mg once daily x 14 days</li> <li>Treatment B = RBT 300 mg once daily + CAB 30 mg once daily x 14 days</li> </ul> |
| Interim<br>Analysis | No interim analysis will be performed. |

## 2.4. Statistical Hypotheses

No formal hypothesis will be tested. This study is designed to estimate the drug-interaction effect of RBT on CAB PK parameters. An estimation approach will be used to evaluate the effect of RBT on CAB PK. Point estimates and corresponding 90% confidence intervals (CIs) will be constructed for the comparisons of interest (test:reference).

### 3. PLANNED ANALYSIS

## 3.1. Interim Analyses

• No interim analysis will be performed.

## 3.2. Final Analyses

Final analyses will be performed after the completion of the study, following sequential steps and final database authorization:

- 1. All subjects have completed the study as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.
- 3. All criteria for unblinding the randomisation codes have been met.
- 4. Randomisation codes have been distributed according to RandAll NG procedures.

### 4. ANALYSIS POPULATIONS

| Population Definition / Criteria | | Analyses Evaluated |
|---|---|---|
| Screening<br>Population | All subjects who sign the consent form will be included in this population. | Screening population<br>listing and summary |
| Safety<br>Population | All subjects who enrol in the study and receive at least one dose of study drug will be included in the Safety Population. | <ul><li>Study Population</li><li>Safety</li></ul> |
| PK<br>Concentration<br>Population | The CAB PK Concentration Population will include all subjects who undergo plasma PK sampling and have evaluable PK assay results. | PK concentration<br>listing, and individual<br>concentration plot |
| PK Parameter<br>Population | The PK Parameter Population will include all subjects who have evaluable PK parameters. Data from subjects who vomit within 4 hours of study drug administration will not be considered as evaluable. | PK parameter listing,<br>and plotting |
| PK Summary<br>Population | The CAB PK Summary Population for this study will include subjects who have CAB PK parameter estimates from both serial PK sampling time periods 1 and 2. These populations will be used for the concentration and PK parameters summary figures and tables and for the statistical analysis of PK parameter data | <ul> <li>PK concentrations<br/>and summary table<br/>and summary figures</li> <li>PK Parameter<br/>Summary table</li> <li>Statistical analysis of<br/>parameter data</li> </ul> |

### NOTES:

• Please refer to Appendix 11 which details the population to be used for each display being generated.

### 4.1. Protocol Deviations

Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, subject management or subject assessment) will be listed.

- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to unblinding and freezing the database to ensure all important deviations and deviations which may lead to exclusion from the PK analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 2 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 2 Overview of Appendices

| Section | Component |
|---|---|
| Section 10.1 | Appendix 1: Protocol Deviation Management |
| Section 10.2 | Appendix 2: Data Management |
| Section 10.3 | Appendix 3: Time & Events |
| Section 10.4 | Appendix 4: Treatment States and Phases |
| Section 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| Section 10.6 | Appendix 6: Derived and Transformed Data |
| Section 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| Section 10.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 10.9 | Appendix 9: Model Checking and Diagnostics for Statistical Analyses. |
| Section 10.10 | Appendix 10: Abbreviations and Trade Marks |
| Section 10.11 | Appendix 11: List of Data Displays |
| Section 10.12 | Appendix 12: Example Mock Shells for Data Displays |

### 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Analyses

The study population analyses will be based on the "Safety" population, unless otherwise specified.

Table 3 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

 Table 3
 Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | | |
|---|---|---|---|
| | Figure | Table | Listing |
| <b>Study Population</b> | | | |
| Analysis Population Summary | | Y | |
| <b>Subject Disposition</b> | | | |
| Subject Disposition | | Y | Y |

| Display Type | Data 1 | Displays Gen | erated |
|---|---|---|---|
| | Figure | Table | Listing |
| Protocol Deviations | | Y | Y |
| Inclusion and Exclusion Criteria Deviations | | | Y |
| Demography | | | |
| Demographics Characteristics | | Y | Y |
| Race & Racial Combinations | | Y | Y |
| Age Group Breakdown for Trial | | Y | |
| Others | | | |
| Concomitant Medication | | $Y^1$ | Y |
| Genetic sample collection | | | Y |
| Random codes | | | Y |
| Treatment non-compliance | | | Y |
| Screening information | | Y <sup>2</sup> | Y <sup>3</sup> |

### NOTES:

- Y = Yes display generated.
- 1. Conditional display, if data contains more than 10 records.
- 2. Screening population.
- 3. All screen failures

## 7. PRIMARY STATISTICAL ANALYSES

## 7.1. Pharmacokinetic Analyses

The reconciliation of the PK Case Report Form (CRF) and SMS2000 data will be performed by Data Management, QSci at GlaxoSmithKline.

The merge of PK concentration data, randomization and CRF data will be performed. The analysis PK concentration dataset and WinNonLin files will be created by statistics and programming, under the direct auspices of statistics and programming, Quantitative Sciences (QSci), GlaxoSmithKline.

Derivation of pharmacokinetic parameters will be performed under the direct auspices of Clinical Pharmacology Modelling & Simulation (CPMS), QSci, GlaxoSmithKline.

Statistical Analysis of pharmacokinetic parameters will be performed by statistics and programming under the direct auspices of statistics and programming, QSci, GlaxoSmithKline.

### 7.1.1. Overview of Planned Pharmacokinetic Analyses

The pharmacokinetic (PK) analyses will be based on the PK Concentration, PK Parameter, or PK Summary populations where it is specified.

Table 4 provides an overview of the planned analyses, with full details being presented in Appendix 11: List of Data Displays.

Table 4 Overview of Planned Pharmacokinetic Analyses

| Endpoints | Ur | itrans | formed | Log <sub>e</sub> -Transformed | | | | |
|---|---|---|---|---|---|---|---|---|
| | Summa | ary | Indiv | idual | Summ | ary | Individual | |
| | F | T | F | L | F | T | F | L |
| Plasma Drug Concentrations | Y [1] [2] | Y | Y [1] | Y | Y [1] [2] | | Y [1] | |
| Derived PK Parameters | | Y | $Y^{[3]}$ | Y | | Y | $Y^{[3]}$ | |
| Statistical Analysis PK Parameters | | | | | Y <sup>[4]</sup> | Y | | Y <sup>[5]</sup> |

### NOTES:

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TF related to any summaries (descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- Tmax is not log transformed.
- 1. Linear and Semi-Log plots will be created on the same display.
- 2. Mean (+SD) and Median plots will be generated.
- 3. Comparative Plot of Individual CAB Plasma PK Parameter vs treatments on linear and semi-log scale
- 4. Geometric Mean Treatment Ratio and 90% CI of CAB Plasma PK Parameters will be generated.
- 5. Supportive SAS Output from Statistical Analysis of Loge-transformed CAB Plasma PK Parameters

### 7.1.2. Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Process & Standards).

### 7.1.3. Pharmacokinetic Parameters

PK analyses will be the responsibility of the CPMS department within GSK or their designee. Plasma CAB concentration-time data will be analyzed by non-compartmental methods according to current working practices and using Phoenix WinNonlin 6.3 or higher. Calculations will be based on the actual sampling times recorded during the study and based on nominal sampling times. From the plasma concentration-time data, the following PK parameters will be determined, as data permit: Cmax, Tmax,  $C\tau$ , t1/2,  $AUC(0-\tau)$  and CL/F.

Statistics and Programming group will calculate the individual ratios for Cmax,  $C\tau$  and  $AUC(0-\tau)$ .

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Process & Standards).

Non-compartmental analysis will be performed in accordance with GSK PK Guidance document GUI 51487.

Refer Appendix 7 Section 10.7.2.2 for handling of PK Concentration data.

Table 5 Derived Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-τ) | Area under the plasma concentration-time curve at the end of the dosing |
| | interval will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental |
| | trapezoid. |
| Cmax | Maximum observed concentration, determined directly from the |
| | concentration-time data. |
| Сτ | Plasma concentration at the end of the dosing interval |
| Tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| t1/2 | Apparent terminal half-life will be calculated as: $t\frac{1}{2} = \ln 2 / \text{Lambda}_z$ |
| | (NOTE: Lambda_z is the terminal phase rate constant). |
| CL/F | The apparent oral clearance (CL/F) will be calculated as CL/F = |
| | Dose/AUC(0-τ) |

PK parameters that have mass in the units should be reported in μg/mL and h•μg/mL for CAB. CL/F should be reported in units of L/h.

### 7.2. Statistical Analysis of Pharmacokinetic Parameters

All PK data will be stored in the Archives, GlaxoSmithKline R& D. Statistical analyses of the PK parameter data will be the responsibility of Clinical Statistics, GlaxoSmithKline or their designee.

For each of the parameters Cmax,  $C\tau$ ,  $AUC(0-\tau)$ , t1/2 and CL/F, if data permit, the following summary statistics will be calculated and tabulated by treatment:

- Untransformed Data: N, n, arithmetic mean, SD, median, minimum, maximum and %CV.
- **Log**<sub>e</sub>-transformed Data: Geometric mean, 95% CI for the geometric mean, SD of log<sub>e</sub>-transformed data and %CVb

For Tmax , the summary statistics specified for untransformed data above will be generated.

### **Primary and Secondary Comparisons of Interest**

| | CAB<br>PK Parameter | Test | Reference | Assessment |
|---|---|---|---|---|
| Primary | Cmax and AUC(0-τ) | Treatment B: RBT+CAB | Treatment A: CAB | Interaction |
| Secondary | Cτ, t1/2 and CL/F | Treatment B: RBT+CAB | Treatment A: CAB | Interaction |

The PK parameters for CAB (except  $T_{max}$ ) will be  $log_e$ -transformed and separately analyzed using a mixed effects model. Analysis of variance (ANOVA), considering treatment as fixed effect and subject will be treated as a random effect in the model, will

be performed using SAS Mixed Linear Models procedure to evaluate the effect of RBT on CAB PK parameters:  $AUC(0-\tau)$  and Cmax. Similar model will be applied for secondary endpoints:  $C\tau$ , t1/2 and CL/F. Point estimates and their associated 90% CIs will be constructed for the differences in PK parameter values between RBT+CAB and CAB alone for the treatment comparisons. The point estimates and their associated 90% CIs will then be back-transformed to provide point estimates and 90% CIs for the ratios of PK parameters between test and reference treatments.

Estimates of within-subject variability for Cmax,  $C\tau$ , t1/2,  $AUC(0-\tau)$  and CL/F will be provided, where  $CVw(\%) = SQRT(exp(MSE) - 1) \times 100$  and MSE is the residual mean squared error from the model. CVw represents a pooled measure of within-subject variability across the treatments CAB and RBT+CAB.

Pre-dose concentrations collected between Days 13-14 and Days 26-28 will be listed with PK concentration profiles and summarized by Day/Time. To assess for achievement of steady-state of CAB when CAB is given with RBT, Analysis of variance (ANOVA), considering DAY as fixed effect and subject as a random effect in the model, will be performed using SAS Mixed Linear Model on the pre-dose concentration between Days. The estimated slope and 90% CI will be presented for models included 2 days (Days 13-14, 27-28) or 3 days (Days 26-28) pre-dose concentrations.

Comparative Plot of Individual subject CAB Plasma PK Parameter Versus Treatment will be generated.

Individual and box plots of Pre-dose concentration of Day 13-14 and Days 26-28 will be generated.

Plots will also be provided showing the adjusted geometric mean ratio of test to reference treatment for Cmax,  $C\tau$ , AUC(0- $\tau$ ), t1/2 and CL/F with 90% CIs.

The SAS output from the statistical models will be included in a listing of supportive SAS output.

## 8. SECONDARY STATISTICAL ANALYSES

### 8.1. Safety Analyses

### 8.1.1. Overview of Planned Analyses

The safety analyses will be based on the Safety population, unless otherwise specified.

Table 6 provides an overview of the planned analyses, with full details of data displays being presented in Appendix 11: List of Data Displays.

Table 6 Overview of Planned Safety Analyses

| Endpoint | | Abs | olute | | Ch | ange fr | om Base | eline |
|---|---|---|---|---|---|---|---|---|
| | Sum | mary | Indi | vidual | Sum | ımary | Indiv | idual |
| | T | F | F | L | T | F | F | L |
| Exposure | | | | | | | | |
| Exposure | Y | | | Y | | | | |
| Adverse Events | | | | | | | | |
| All AE's | Y | | | Y | | | | |
| Serious AE's | | | | Y | | | | |
| Drug Related AEs | Y | | | $Y^1$ | | | | |
| Withdrawal AE's | Y | | | Y | | | | |
| Relationship Between System | | | | Y | | | | |
| Organ Class and Verbatim Text | | | | | | | | |
| Liver Event | | | | Y | | | | |
| Laboratory Values | | | | | | | | |
| Clinical Chemistry | Y | | | $Y^2$ | | | | |
| Hematology | Y | | | $Y^2$ | | | | |
| Clinical Lab Reference Ranges | | | | Y | | | | |
| Treatment Emergent Toxicity | Y | | | | | | | |
| Grade | | | | | | | | |
| Urinalysis | Y | | | Y | | | | |
| ECG's | | | | | | | | |
| ECG Findings | Y | | | Y | | | | |
| ECG Values | Y | | | $Y^2$ | Y | | | |
| Category of QTc Data | Y | | | | Y | | | |
| ECG Values Outside the PCI | | | | Y | | | | |
| Range | | | | | | | | |
| Vital Signs | | | | | | | | |
| Vitals Values | Y | | | $Y^2$ | Y | | | |
| Vital Signs Measurements | | | | Y | | | | |
| Outside the PCI Range | | | | | | | | |

### **NOTES:**

- T = Table, F = Figures, L = Listings, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data
- Individual = Represents FL related to any displays of individual subject observed raw data.
  - 1: Part of all AEs listing
  - 2: Listing will include toxicity grade or flag for H/L if out of normal range

### 9. REFERENCES

GlaxoSmithKline Document Number 2016N269788\_00: Phase I, single-center, open label, fixed-sequence cross-over study to evaluate the effect of rifabutin on the pharmacokinetics of oral cabotegravir in healthy subjects. Effective Date: 23-FEB-2017

GlaxoSmithKline Document Number 2016N269788\_01: Phase I, single-center, open label, fixed-sequence cross-over study to evaluate the effect of rifabutin on the pharmacokinetics of oral cabotegravir in healthy subjects Effective Date: 13-APR-2107

GlaxoSmithKline Document Number 2016N269788\_02: Phase I, single-center, open label, fixed-sequence cross-over study to evaluate the effect of rifabutin on the pharmacokinetics of oral cabotegravir in healthy subjects Effective Date: 29-Jun-2017

## 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 10.1 | Appendix 1: Protocol Deviation Management |
| RAP Section 5 Conventions | : General Considerations for Data Analyses & Data Handling |
| Section 10.2 | Appendix 2: Data Management |
| Section 10.3 | Appendix 3: Time and Events |
| Section 10.4 | Appendix 4: Treatment States & Phases |
| Section 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.6 | Appendix 6: Derived and Transformed Data |
| | General |
| | Study Population |
| | • Safety |
| | Pharmacokinetic |
| Section 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | General |
| | Study Population & Safety |
| Section 10.8 | Appendix 8: Values of Potential Clinical Importance |
| | Laboratory Values |
| | • ECG |
| | Vital Signs |
| Section 10.9 | Appendix 9: Model Specifications for Statistical Analyses |
| Other RAP A | ppendices |
| Section 10.10 | Appendix 10: Abbreviations & Trade Marks |
| Section 10.11 | Appendix 11: List of Data Displays |
| Section 10.12 | Appendix 12: Example Mock Shells for Data Displays |

## 10.1. Appendix 1: Protocol Deviation Management

## **10.1.1.** Exclusions from PK Parameter Summary Population

All protocol deviations will be reviewed, and only the important deviations will be listed and summarized. Some subjects may be excluded from analysis due to protocol deviations. A subject meeting any of the following criteria will be excluded from the PK Parameter Summary Population:

| Number | Exclusion Description |
|---|---|
| 01 | Failure of any inclusion/exclusion criteria, but subject is still enrolled |
| 02 | A subject with emesis occurring within 4 hours of the dose on Day 14 or Day 28 |
| 03 | A subject who does not have evaluable PK parameters from both periods |
| 04 | A subject who has not dosed correctly on the days for PK collections |

## 10.2. Appendix 2: Data Management

### 10.2.1. Data Format and Process

| Data Type | Source | Format of Data | Planned Date of Final File | Responsibi lity |
|---|---|---|---|---|
| Safety | PIMS>SI data | SI>STDM | DBF | Accenture |
| PK<br>Concentration | SMS2000 data file | dat file | DBF | BIB/BESM |
| PK<br>Concentration<br>(ADPC),<br>WNL File | PK concentration data (SDTM PC), exposure (EX) and demography (DM) datasets <sup>2</sup> | ADaM, CSV<br>file | DBF + 5 Days <sup>1</sup> | QSci |
| PK<br>Parameters | WNL file | CSV file | PK<br>Concentration,<br>WNL file + 10<br>Days | CPMS |

<sup>1.</sup> Provided SDTM PC, EX and DM are in time and clean

<sup>2.</sup> PK concentration data is released via SMS2000 by Bioanalysis, Immunogenicity and Biomarkers (BIB)/Bioanalytical External Study Monitors (BESM) and the SDTM PC contains date/times and PK sample ID

# 10.3. Appendix 3: Time & Events

## 10.3.1. Protocol Defined Time & Events

| Procedure | Screen <sup>1</sup> | Day<br>-1 | | Treatment Period 1<br>Day | | | | | | | | | | | | | Treatment Period 2 Day | | | | | | | | | | | | | | Early<br>Withdrawal<br>/ Follow-up<br>~10-14<br>days | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | _ | 2 | ယ | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 212 | 22 | 23 | 24 | 25 | <b>26</b> <sup>2</sup> | 27 | 28 | 29 | |
| Informed consent | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Inclusion and exclusion criteria | Х | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Demography | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Full physical exam <sup>3</sup> | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Brief physical exam <sup>3</sup> | | Х | | | | | | | | | | | | | | Х | | | | | | | Х | | | | | | | Х | | X <sup>4</sup> |
| Medical/medicatio<br>n/drug/alcohol<br>history | Х | Х | | | | | | | | | | | | | | Х | | | | | | | Х | | | | | | | | | |
| Pregnancy test 5 | Χ | Χ | | | | | | | | | | | | | | Χ | | | | | | | | | | | | | Χ | | | Χ |
| FSH and estradiol (if needed) | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| TB, HIV, Hep B,<br>Hep C screen | Х | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Drug/Alcohol<br>screen | Х | Х | | | | | | | | | | | | | Χ | | | | | | | | | | | | | | Χ | | | |

| Procedure | Screen <sup>1</sup> | Day<br>-1 | | Treatment Period 1<br>Day | | | | | | | | | | | | | | Treatment Period 2<br>Day | | | | | | | | | | | | | | Early<br>Withdrawal<br>/ Follow-up<br>~10-14<br>days |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 1 | 2 | ယ | 4 | 5 | 6 | 7 | ∞ | 9 | 10 | 1 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | <b>21</b> <sup>2</sup> | 22 | 23 | 24 | 25 | <b>26</b> <sup>2</sup> | 27 | 28 | 29 | |
| Safety Laboratory assessments | Х | Х | | | | | | | | | | | | | Χ | | | | | | | | Х | | | | | | Х | | | Х |
| 12-lead ECG <sup>6</sup> | Χ | | Χ | | | | | | | | | | | | | Χ | | | | | | | | | | | | | | Χ | | Х |
| Vital signs<br>(Including<br>Temperature) <sup>6</sup> | Х | | Х | | | | | | | | | | | | | Х | | | | | | | Х | | | | | | | Х | | Х |
| Administer CAB<br>30 mg once daily <sup>7</sup> | | | Х | Χ | Х | Χ | Х | Χ | Χ | Χ | Х | Х | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Х | Х | Χ | Χ | Х | Χ | Х | Χ | | |
| Administer RBT<br>300 mg once<br>daily <sup>7</sup> | | | | | | | | | | | | | | | | | Х | Χ | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | |
| Dispense CAB8 | | | Χ | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Dispense<br>CAB <sup>9</sup> and RBT <sup>10</sup> | | | | | | | | | | | | | | | | | Х | | | | | | | | | | | | | | | |
| Pharmacokinetic Sampling <sup>11</sup> | | | | | | | | | | | | | | | Х | X | -X | | | | | | | | | | | Χ | Χ | X<br>X | | |
| Admit to Unit | | Χ | | | | | | | | | | | | | Χ | | | | | | | | | | | | | | Χ | | | |
| Discharge from<br>Unit | | | Χ | | | | | | | | | | | | | | Χ | | | | | | | | | | | | | | X | |
| Outpatient Visit | Χ | | | | | | | | | | | | | | | | | | | | | | Χ | | | | | Χ | | | | Χ |

| Procedure | Screen <sup>1</sup> | Day<br>-1 | | Treatment Period 1<br>Day | | | | | | Treatment Period 2<br>Day | | | | | | | Early<br>Withdrawal<br>/ Follow-up<br>~10-14<br>days | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 | 19 | 20 | 212 | 22 | 23 | 24 | 25 | <b>26</b> <sup>2</sup> | 27 | 28 | 29 | |
| Drug<br>accountability | | | | | | | | | | | | | | | Х | | | | | | | | Х | | | | | Х | Х | | | |
| Genetic sample <sup>12</sup> | | | <b>←</b> | -=== | === | :=== | ===: | ==== | === | === | ===: | ==== | :===: | ==== | ==== | ===== | ==== | ===: | ==== | ==== | ==== | ==== | ==== | :===: | ==== | :===: | ==== | ===: | ==== | ==== | ==== | ====→ |
| SAE Review | <b>←====</b> | ===== | ==== | ==== | ==== | | === | ===: | ==== | === | === | ==== | === | ==== | === | ===== | ==== | :=== | ==== | ===: | ==== | ==== | === | === | ==== | === | ==== | === | ==== | ===: | ==== | ===== <del>)</del> |
| AE Review | | | <b>+</b> | -=== | === | === | === | ==== | === | === | === | ==== | === | ==== | ==== | | ==== | === | ==== | ==== | === | ==== | ==== | === | ==== | === | ==== | === | ==== | ==== | === | ====> |
| Concomitant medication review | | | + | -=== | | :===: | ===: | ==== | === | === | ===: | ==== | ===: | ==== | ==== | ===== | ==== | ===: | ==== | ==== | === | ==== | ==== | ===: | ==== | ===: | ==== | ===: | ==== | ==== | ==== | ====→ |

- 1. Screening must be performed within 30 days prior to receiving the dose of CAB on Day 1.
- 2. Day 21 and Day 26 is an outpatient visit.
- 3. An ocular assessment will be performed only for subjects who experience eye symptoms.
- 4. A brief symptom directed physical exam will be completed as needed.
- 5. A serum pregnancy test will be performed at the screening visit and a urine pregnancy test at all other time points specified.
- 6. Duplicate ECG, BP, and HR assessments will be conducted pre-dose on Day 1. Single measurements will be collected at all other time points.
- 7. Study medication will be administered with 240 mL of water within the unit on Days 1, 13, 14, 15, 21, 26, 27, and 28. Dosing on non-PK days may be with or without food, but dosing on serial PK days (Day 14 in Period 1 and Day 28 in Period 2) must be after an overnight fast of at least 6 hours, and no food will be allowed for 4 hours after dosing on these serial PK days.
- 8. Dispense the bottle of CAB tablets to the subject on Day 1 to receive CAB dosing at home on Days 2 to 12 in Period 1
- 9. Dispense the bottle of CAB tablets to the subject on Day 15 to receive CAB dosing at home on Days 16 to 20 and Days 22 to 25 in Period 2; dosing on Day 21, 26, 27, and 28 is in the unit.
- 10. Dispense the bottle of RBT capsules to the subject on Day 15 to receive RBT dosing at home on Days 16 to 20 and Days 22 to 25 in Period 2; dosing on Day 21, 26, 27, and 28 is in the unit.
- 11. Plasma PK samples (2 mL of blood per sample) will be collected to measure CAB at the following time points: Period 1: predose (within 15 minutes prior to dose) on Day 13; and pre-dose (within 15 minutes prior to dose), 1, 2, 3, 4, 8, 12, and 24 hours after CAB dosing on Day 14. Period 2: pre-dose (within 15 minutes prior to dose) on Days 26 and 27 and pre-dose (within 15 minutes prior to dose) on Day 28 and, 1, 2, 3, 4, 8, 12, and 24 hours after CAB +RBT dosing on Day 28.
- 12. It is recommended that the Pharmacogenetic sample be collected on Day 1, but it may be collected at any time following administration of investigational product.

## 10.4. Appendix 4: Treatment States and Phases

### 10.4.1. Treatment State and Study Phases

Assessments and events will be classified according to the time of occurrence relative to study visit or the start and/or stop date/time of the study treatment.

| Treatment<br>State | Study Phase |
|---|---|
| Pre-Treatment | Screening assessments collected prior to the Day 1 visit |
| On-Treatment | Period 1 and Period 2 |
| Follow-up | Follow-up Visit |

## 10.4.1.1. Treatment States for AE, SAE and Concomitant Medications Data

| Treatment<br>State | Definition |
|---|---|
| Screening | AE(SAE or conmed) Start Date/Time < Study Treatment Start Date/Time. Based on the protocol, these AEs and concomitant medications prior to dosing will not be collected in database, and only record in the source document, but SAE will be captured on the dataset |
| Treatment A | If AE (SAE or conmed) onset date/time is on or after Period 1 treatment start date/time & before Period 2 treatment date/time Study Period 1 Treatment Start Date/Time ≤ AE Start Date/Time < Study Period 2 Treatment Date/Time] |
| Treatment B | If AE (SAE or conmed) onset date/time is on or after Period 2 treatment start date/time & before Study Conclusion date/time Study Period 2 Treatment Start Date/Time ≤ AE Start Date/Time < Study follow-up visit Date/Time] |
| Follow-up | All unsolved AEs (SAE or conmed) during the follow-up will be associated with the treatment from Period 2, and no AEs (SAE or conmed) will be report under the follow-up |
| Onset Time<br>Since First<br>Dose<br>(Days) | If Treatment Start Date/Time > AE Onset Date/Time = AE Onset Date - Treatment Start Date If Treatment Start Date/Time ≤ AE Onset Date/Time = AE Onset Date - Treatment Start Date +1 Missing otherwise |
| Duration<br>(Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on eCRF |

### **NOTES:**

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

## 10.4.1.2. Reporting Other Safety Data

All of other safety measurements will be associated and summarized for each visit based on the CRF as the following:

| Visit | Time Slices Definition |
|-----------|--------------------------------|
| Screening | Screen |
| Period 1 | Day -1, Period 1 Days 1-Day 14 |
| Period 2 | Period 2, Days 15-28 |
| Follow-up | Follow-up |

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

## 10.5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | |
|---|---|---|
| | RandAll NG | Data Displays for<br>Reporting |
| Code | Description and Footnotes for the Displays | Description |
| A | CAB 30 mg once daily x 14 days | CAB 30mg |
| В | RBT 300 mg once daily + CAB 30 mg once daily x 14 days | RBT 300mg + CAB<br>30mg |

### 10.5.2. Baseline Definition & Derivations

### 10.5.2.1. Baseline Definitions

For all endpoints (except as noted in the table) the baseline value will be the latest predose assessment.

Table 7 Baseline Definitions

| Danamatan | Study Asses | ssments C<br>Baseline | Baseline Used in | |
|---|---|---|---|---|
| Parameter | Screening | Day -1 | Day 1<br>(Pre-Dose) | Data Display |
| Safety | | | | |
| Labs | X | X | | Day -1 |
| ECG | | | X | Day 1 (Pre-Dose) |
| Vital Signs (blood pressure, and pulse rate) | X | | X | Day 1 (Pre-Dose) |

## 10.5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline |

### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.5.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

## 10.5.3. Reporting Process & Standards

| Reporting Process | |
|---|---|
| Software | |
| The currently supported versions of SAS and S-Plus software will be used. | |
| Reporting Area | |
| HARP Server | : US1SALX00259-HARP PROD-US |
| HARP Area | : \ARPROD\GSK1265744\mid205712\Final |
| QC Spreadsheet | : \ARWORK\GSK1265744\mid205712\Final\Documents |
| <b>Analysis Datasets</b> | |
| <ul> <li>Analysis datasets will be created according to Clinical Data Interchange<br/>Standards Consortium (CDISC) standards (SDTM IG Version 3.1.3 or higher<br/>vision &amp; Analysis Data Model (ADaM) Implementation Guide (ADaM IG)<br/>Version 1.1 or higher dataset standards)</li> </ul> | |
| Generation of Rich Text Format (RTF) Files | |
| RTF files will be generated for Safety summary displays. | |

### **Reporting Standard**

### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - o 4.03 to 4.23: General Principles
  - o 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - o 7.01 to 7.13: Principles Related to Graphics

### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - o Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| Reporting Standard | |
|---|---|
| Descriptive Summary | Statistics |
| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharma | cokinetic Concentration Data |
| Descriptive Summary<br>Statistics | Refer to IDSL Statistical Principle 6.06.1 Assign zero to NQ values (Refer to GUI_51487 for further details) |
| Reporting of Pharma | cokinetic Parameters |
| Descriptive Summary Statistics. (Un-Transformed) Descriptive Summary Statistics. (Loge Transformed) | <ul> <li>N, n, arithmetic mean, 95% confidence interval (CI) for the arithmetic mean, SD, median, minimum, maximum and CV(%)</li> <li>CV(%)=(SD/mean)*100</li> <li>N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between-subject geometric coefficient of variation (CVb (%)) will be reported.</li> <li>Geometric mean = exp (mean on loge scale)</li> <li>CVb (%) = √ (exp(SD²) - 1) * 100 [NOTE: SD = SD of loge transformed data]</li> </ul> |
| Parameters Not<br>Being Log <sub>e</sub><br>Transformed | Tmax |
| Listings | Include PK Parameters: Cmax, Tmax, $C\tau$ , $AUC(0-\tau)$ , $t1/2$ and $CL/F$ . |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

## 10.6. Appendix 6: Derived and Transformed Data

### 10.6.1. **General**

### **Multiple Measurements at One Time Point**

• Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.

### **Study Day**

- Calculated as the number of days from Treatment start date :
  - Ref Date = Missing
- $\rightarrow$  Study Day = Missing
- Ref Date < Treatment start Date → Study Day = Ref Date Treatment start Date
- Ref Data ≥ Treatment start Date → Study Day = (Ref Date Treatment start Date) + 1

## 10.6.2. Study Population

### **Demographics**

### Age

- GSK standard IDSL algorithms will be used for calculating age using date of the screening visit relative to birth date, where birth date is imputed as:
  - Any subject with a missing date and month will have this imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / [Height (m)]<sup>2</sup>

### **Extent of Exposure**

Number of days of exposure to study drug will be calculated based on the formula:
 Duration of Exposure in Days = Treatment Stop Date - (Treatment Start Date) + 1

### 10.6.3. Safety

### **ECG Parameters**

### **RR** Interval

• IF RR interval (msec) is not provided directly, then RR can be derived as:

[1] If QTcB is machine read & QTcF is not provided, then:

$$RR = [(QT/QTcB)^{(2)}]*1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = [(QT/QTcF)^{3}]*1000$$

### **Corrected QT Intervals**

• When not entered directly in the eCRF, corrected QT intervals using Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.

• IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

## **Laboratory Parameters**

• If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.

• Example 1: 2 Significant Digits = < x becomes x - 0.01

• Example 2: 1 Significant Digit = '> x' becomes x + 0.1

• Example 3: 0 Significant Digits = '< x' becomes x – 1

# 10.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

## 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | All subjects who withdraw prematurely from the study/study drug will be documented, listed with the reason for their withdrawal recorded in the final Clinical Pharmacology Study Report (CPSR). |

## 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing PK and safety data will not be imputed |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented and flagged in the dataset and listing along with the reason for exclusion in the clinical study report. |

## 10.7.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: O Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 4: Treatment States and Phases. Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used. Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing. |

## 10.7.2.2. Handling of PK Concentration Data

| Element | Reporting Detail |
|---|---|
| General | If a PK sample in a profile is 'no result', 'no sample received', or 'insufficient sample', data will be set as missing. No imputation will be applied. |

## 10.8. Appendix 8: Values of Potential Clinical Importance

### 10.8.1. Laboratory Values

Division of AIDS (DAIDS, Version 2.0, November 2014) AE grade 2 and above of lab abnormalities will be listed by subject, period/treatment, visit, and actual date and time.

Statistics and Programming group will use this version to add toxicity grades values in the ADAM dataset.

### 10.8.2. ECG

### **ECG Values of Potential Clinical Importance (Healthy Volunteers)**

| ECG Parameter | Potential Clinical Importance Range (PCI) | Unit |
|---|---|---|
| Absolute QTc Interval | >450 | msec |
| Increase from baseline QTc | >60 | msec |
| PR Interval | <110 and >220 | msec |
| QRS Interval | <75 and >110 | msec |

## 10.8.3. Vital Signs

## **Vital Signs Values of Potential Clinical Importance (Healthy Volunteers)**

| Parameter | Potential Clinical Importance Range (PCI) | Unit |
|--------------------------|-------------------------------------------|------|
| Systolic Blood Pressure | <85 and >160 | mmHg |
| Diastolic Blood Pressure | <45 and >100 | mmHg |
| Heart Rate | <40 and >110 | bpm |

## 10.9. Appendix 9: Model Specifications for Statistical Analysis

## 10.9.1. Statistical Analysis Assumptions and Model Specifications

| <b>Endpoint(s)</b> | Cmax, $C\tau$ , AUC(0- $\tau$ ), t1/2 and CL/F, if data permitted |
|---|---|
| Analysis | Linear Mixed Model |

### **Specifications:**

- For the Linear Mixed Model, model assumptions will be PK parameter following lognormal distribution.
- For drug-drug interaction assessment, an example of SAS code is included here.

• An example of SAS code to assess achievement of steady-state is included here.

```
Proc Mixed;
   by dose;
   where day in (13,14);
   class subject;
   model logC0 = day/ddfm=kr cl alpha=0.1 solution;
   random intercept/subject=subject type=un solution;
   make 'solutionf' output=stat;
run;
```

repeat for Days 26,27,28 and Days 27,28

# 10.10. Appendix 10 - Abbreviations & Trade Marks

## 10.10.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| ADaM IG | Analysis Data Model Implementation Guide |
| AE | Adverse Event |
| ANOVA | Analysis of Variance |
| AUC | Area under concentration-time curve |
| AUC(0-τ) | Area under the concentration-time curve over one dosing interval |
| BESM | Bioanalytical External Study Monitors |
| BIB | Bioanalysis, Immunogenicity and Biomarkers |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CL/F | The apparent oral clearance |
| Cmax | Maximum observed concentration |
| СР | Clinical Programming |
| CPMS | Clinical Pharmacology Modelling & Simulation |
| CPSSO | Clinical Pharmacology Sciences and Study Operations |
| CRF | Case record form |
| CS | Clinical Statistics |
| Ct | Concentration at the end of the dosing interval |
| CV | Coefficient of Variation |
| CVb/CVw | Coefficient of Variation (Between)/Coefficient of Variation (Within) |
| DAIDS | Division of Acquired Immune Deficiency Syndrome |
| DBF | Database Freeze |
| DBR | Database Release |
| GSK | GlaxoSmithKline |
| HARP | Harmonized Analysis and Reporting Process |
| IDSL | Integrated Data Standards Library |
| LLQ | Lower limit of quantification |
| NC | Not Calculable |
| NQ | Non-quantifiable concentration measured as below LLQ |
| PK | Pharmacokinetic |
| QSci | Quantitative Sciences |
| RAP | Reporting and Analysis Plan |
| RBT | Rifabutin |
| RTF | Rich Text Format |
| SAS | Statistical Analysis System |
| SD | Standard deviation |
| SDTM | Study Data Tabulation Model |
| SRP | Statistics Resourcing and Programming |
| t½ | Terminal phase half-life |
| Tmax | Time of occurrence of Cmax |
## 10.10.2. Trademarks

| Trademarks of ViiV Healthcare | Trademarks not owned by ViiV<br>Healthcare |
|-------------------------------|--------------------------------------------|
| NONE | Mycobutin |
| | SAS |
| | WinNonlin |

## 10.11. Appendix 11: List of Data Displays

### 10.11.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|------------------|------------|------------|
| Study Population | 1.1 to 1.n | N/A |
| Safety | 2.1 to 2.n | N/A |
| Pharmacokinetic | 3.1 to 3.n | 3.1 to 3.n |
| Section | Lis | tings |
| ICH Listings | 1 : | to x |
| Other Listings | x+1 | to y |

### 10.11.2. Mock Example Referencing

All displays will be provided with an example from previous CAB studies LAI117010 and LAI117011 or mock examples are provided.

# 10.11.3. Study Population Tables

| Study | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | <b>Programming Notes</b> | Deliverable [Priority] |
| Subjec | ct Disposition | | | | |
| 1.1. | Safety | LAI117010/ Table 1.1 | Summary of Analysis Populations | by Overall | SAC |
| 1.2. | Safety | LAI117010/ Table 1.2 | Summary of End of Study Record by Treatment and Overall | By subject and treatment | SAC |
| 1.3. | Safety | LAI117010/ Table 1.3 | Listing of End of Study Record | By subject | SAC |
| Demog | graphics and E | nrolment Information | | | |
| 1.4. | Safety | LAI117010/ Table 1.5 | Summary of Demographic characteristics | Include BMI, Race detail | SAC |
| 1.5. | Safety | LAI117010/ Table 1.6 | Summary of Race for Safety Population | By treatment and Overall | SAC |
| 1.6. | Safety | LAI117010/ Table 1.7 | Listing of Concomitant Medication | By Subject. Change from listing to summary if more than 3 pages | SAC |
| 1.7. | Safety | LAI117010/ Table 1.8 | Listing of Genetics Subject Accountability | | SAC |
| 1.8. | Safety | LAI117010/ Table 1.9 | Listing of Treatment Non-Compliance | | SAC |
| 1.9. | Safety | LAI117010/Table 1.10 | Listing of Subjects with Protocol Deviations | | SAC |
| 1.10. | Safety | LAI117010/Table 1.11 | Summary of Screening Information | | SAC |
| 1.11. | Safety | LAI117011/Table 1.11 | Age Group Breakdown for the Trial | For Eudra posting | |

# 10.11.4. Safety Tables

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Adverse l | Events | | | | |
| 2.1. | Safety | LAI117010/ Table 2.1 | Summary of Exposure Data | By subject and treatment | SAC |
| 2.2. | Safety | LAI117010/ Table 2.2 | Relationship of Adverse Event System Organ<br>Classes, Preferred Terms, and Verbatim Text | | SAC |
| 2.3. | Safety | LAI117010/ Table 2.3 | Summary of All Adverse Events by<br>Treatment | | SAC |
| 2.4. | Safety | LAI117010/ Table 2.4 | Summary of Drug-Related Adverse Events by Treatment | | SAC |
| 2.5. | Safety | LAI117010/ Table 2.5 | Listing of Serious Adverse Events | By subject and treatment. | SAC |
| 2.6. | 6. Safety LAI117010/ Table 2.6 | | Listing of Adverse Events Leading to<br>Permanent Discontinuation of Study Drug or<br>Withdrawal from Study | By subject and treatment | SAC |
| Labs | _ | | | | |
| 2.7. | Safety | LAI117010/ Table 2.7 | Listing of Reference Ranges for Clinical Laboratory Tests | | SAC |
| 2.8. | Safety | LAI117010/ Table 2.8 | Summary of Clinical Haematology<br>Laboratory Data by Treatment and Time | | SAC |
| 2.9. | Safety | LAI117010/ Table 2.9 | Summary of Clinical Chemistry Laboratory Data by Treatment and Time | | SAC |
| 2.10. | Safety | LAI117010/ Table 2.10 | Summary of Treatment Emergent Grade 2 or<br>Higher Lab Abnormalities by Treatment | Summary of Treatment<br>Emergent Lab toxicity<br>only. | SAC |
| 2.11. | Safety | LAI117010/ Table 2.11 | Listing of Treatment Emergent Grade 2 or<br>Higher Lab Abnormalities | By subject and treatment | SAC |
| 2.12. | Safety | CP_LB5 | Summary of All Urinalysis Data | | SAC |

| Safety Tab | les | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Signs | } | | | | |
| 2.13. | Safety | LAI117010/ Table 2.13 | Summary of Vital Signs by Treatment and Time | Include BP and HR only. | SAC |
| 2.14. | Safety | LAI117010/ Table 2.14 | Summary of Change from baseline in Vital Signs by Treatment and Time | Include BP and HR only. | SAC |
| 2.15. | Safety | LAI117010/ Table 2.15 | Listing of Vital Signs for Subjects with<br>Abnormalities of Potential Clinical<br>Importance | By subject and treatment | SAC |
| ECGs | | | | | |
| 2.16. | Safety | LAI117010/ Table 2.16 | Summary of ECG Findings | | SAC |
| 2.17. | Safety | LAI117010/ Table 2.17 | Summary of ECG Values by Treatment and Time | | SAC |
| 2.18. | Safety | LAI117010/ Table 2.18 | Summary of Change from Baseline in ECG<br>Values by Treatment and Time | | SAC |
| 2.19. | Safety | LAI117010/ Table 2.19 | Summary of Category of QTc Data by<br>Treatment and Time | | SAC |
| 2.20. | Safety | LAI117010/ Table 2.20 | Summary of Category of QTc Change from Baseline by Treatment and Time | | SAC |
| 2.21. | Safety | LAI117010/ Table 2.21 | Listing of ECG Values for Subjects with<br>Abnormalities of Potential Clinical<br>Importance | By subject and treatment | SAC |
| 2.22. | Safety | LAI117010/ Table 2.22 | Listing of Clinically Significant ECG<br>Abnormalities | List all data for a subject with clinically significant abnormalities | SAC |
| 2.23. | Safety | LAI117011/Table 2.17 | Summary of Serious Adverse Events by<br>Preferred Term Including Drug-related Status<br>and Fatal Status | Eudra posting table | SAC |
| 2.24. | Safety | LAI117011/Table 2.18 | Summary of Non-Serious Adverse Evens by Preferred Term with Occurrences >5% | Eudra posting table | SAC |

| Safety Tables | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | <b>Programming Notes</b> | Deliverable<br>[Priority] |
| 2.25. | Safety | IDSL LIVER5 | Listing of Liver Monitoring and stopping Event Reporting | IDSL standard for liver event | SAC |

#### 10.11.5. Pharmacokinetic Tables

| Pharmac | Pharmacokinetic Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title Pr | | Deliverable<br>[Priority] |
| 3.1. | PK Summary | LAI117010/Table 3.1 | Summary of CAB Plasma Concentration-time Data (unit) by Treatment | Treatments A, B | SAC |
| 3.2. | PK Parameter | LAI117010/Table 3.2 | Listing of Derived Plasma CAB PK Parameters | All parameters with units; | SAC |
| 3.3. | PK Summary | LAI117010/Table 3.3 | Summary of Derived Plasma CAB PK Parameters | All parameters with units | SAC |
| 3.4. | PK Summary | LAI117010/Table 3.4 | Listing of Individual Plasma CAB PK Parameter Treatment Ratios | For Cmax, AUC(0- $\tau$ ), C $\tau$ | SAC |
| Statistica | Statistical Analysis Table | | | | |
| 3.5. | PK Summary | LAI117010/Table 3.5 | Summary of Statistical Analysis of CAB Plasma PK<br>Parameters Comparison | | SAC |
| 3.6. | PK Summary | ITZ112929/Table 11.9 | Summary of Stead-State Assessment | | SAC |

# 10.11.6. Pharmacokinetic Figures

| Pharma | Pharmacokinetic Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID / Example<br>Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| 3.1. | PK Plasma<br>Concentration | LAI117010/ Figure 3.1 | Individual CAB Plasma Concentration-time Plot (Linear and Semi-log) by Subject | Paged by Subject | SAC |
| 3.2. | PK Summary | LAI117010/ Figure 3.2 | Median Plasma CAB Concentration-Time Plots by<br>Treatment (Linear and Semi-Log) | | SAC |
| 3.3. | PK Summary | LAI117010/ Figure 3.3 | Mean Plasma CAB Concentration-Time Plots by<br>Treatment (Linear and Semi-Log) | | SAC |
| 3.4. | PK Summary | LAI117010/ Figure 3.4 | Comparative Plot of Plasma CAB PK Parameters between Treatments | PK_F1 mock up | SAC |
| 3.5. | PK Summary | LAI117010/ Figure 3.5 | Geometric Mean Treatment Ratios and 90% CIs of CAB PK Parameters | PK_F2 mock up | SAC |

## **10.11.7. ICH Listings**

| ICH | ICH Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | <b>Programming Notes</b> | Deliverable [Priority] |
| Rand | Randomisation | | | | |
| 1 | Safety | CP_RA1x (XO) | Listing of Randomized and Actual Treatments | Add randomization date | SAC |
| Subje | ect Disposition | | | | |
| 2 | Screening | ES7 | Listing of Reasons for Screening Failures | Include Age and Sex. Concatenate with Subjid | SAC |
| 3 | Safety | CP_ES10x (XO) | Listing of Reasons for Withdrawal | | SAC |
| 4 | Safety | IE4 (XO) | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC |
| Demo | graphics | | | • | |
| 5 | Safety | DM4 (XO) | Listing of Demographic Characteristics | | SAC |
| 6 | Safety | DM10 (XO) | Listing of Race | | SAC |
| Conc | Concomitant Medication | | | | |
| 7 | Safety | CP_CM4<br>(XO) | Listing of Concomitant Medications by Generic Term | | SAC |
| Expo | sure | | | | |
| 8 | Safety | EX4 (XO) | Listing of Exposure Data | | SAC |

| ICH : | Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | <b>Programming Notes</b> | Deliverable [Priority] |
| Adve | rse Events | | | | |
| 9 | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC |
| 10 | Safety | CP_AE9 (XO) | Listing of All Adverse Events | | SAC |
| LAB | S | | | | |
| 11 | Safety | CP_LB6 (xo) | Listing of Clinical Chemistry | Include all tests, toxicity grades and range flags | SAC |
| 12 | Safety | CP_LB6 (xo) | Listing of Hematology | Include all tests, toxicity grades and range flags | SAC |
| 13 | Safety | UR2b | Listing of Urinalysis Data | | SAC |
| ECG | S | | | | |
| 14 | Safety | CP_EG4 (xo) | Listing of ECG Values of Potential Clinical Importance | | SAC |
| 15 | Safety | CP_EG4 (xo) | Listing of All ECG Values for Subjects with any Value of Potential Clinical Importance | | SAC |
| 16 | Safety | CP_EG6 (xo) | Listing of Abnormal ECG findings | | SAC |
| Vital | Signs | | | | |
| 17 | Safety | CP_VS5 (XO) | Listing of Vital Signs of Potential Clinical Importance | | SAC |
| 18 | Safety | CP_VS5 (XO) | Listing of All Vital Signs for Subjects with any Value of Potential Clinical Importance | | SAC |

## 10.11.8. Non-ICH Listings

| Non- | Non-ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Shell | | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| PK | | | | | |
| 19 | PK Plasma<br>Concentration | pkcl1x | Listing of CAB Plasma Concentration-time Data | | SAC |
| 20 | PK Summary | N/A | SAS Output from Statistical Analysis of Loge-transformed CAB<br>Plasma PK Parameters of Treatment Comparison | | SAC |

## 10.12. Appendix 12: Example Mock Shells for Data Displays

### 10.12.1. Data Display Numbering

The following numbering will be applied for RAP generated displays:

Example : PK\_T1

Protocol: 205712 Page 1 of n

Population : PK Parameter Summary

Table xx.xx

Summary of Statistical Analysis of Log<sub>e</sub>-transformed CAB Plasma Pharmacokinetic Parameters based on Actual Sampling Time

| Parameter | Comparison<br>Test vs Reference | Adjusted (<br>n Test | Geometric Mean<br>n Ref | Ratio<br>(Test/Ref) | 90% Confidence<br>Interval for Ratio | %CVw |
|---|---|---|---|---|---|---|
| Cmax(units) | [Test treatment description] vs<br>[Reference treatment description] | x xx.xx | x xx.xx | x.xxxx | (x.xxxx, x.xxxx) | xx.x |
| AUC(0-τ)(units) | [Test treatment description] vs<br>[Reference treatment description] | x xx.xx | x xx.xx | x.xxxx | (x.xxxx, x.xxxx) | xx.x |
| Cτ(units) [Te | est treatment description] vs<br>[Reference treatment description] | x xx.xx | x xx.xx | x.xxxx | (x.xxxx, x.xxxx) | xx.x |

Example LIVER5

Protocol: XYZ100001 Page 1 of 1
Population: Intent-to-Treat/Safety/Other study specific (Data as of: 30MAY2011)

Tieting

Listing X

Listing of Liver Monitoring/Stopping Event Reporting

| Treatment: Treatment A | | | | | | | |
|---|---|---|---|---|---|---|---|
| Site Id./<br>Unique Subject<br>Id. | Age(YEARS)/<br>Sex/<br>Race Detail | Maximum Status<br>of the Liver<br>Event | Date<br>First<br>Detected/<br>Study Day | Time<br>Since<br>First<br>Dose<br>(days) | Time<br>Since<br>Last<br>Dose<br>(days) | Restart/Re-<br>challenge<br>After<br>Stopping<br>Criteria Was<br>Met | Resolved?/<br>Date<br>resolved |
| PPD | 63/<br>M/<br>WHITE -<br>WHITE/CAUSASIAN/EUROPEAN<br>HERITAGE | LIVER MONITORING<br>CRITERIA | <b>PPD</b> 101 | 101 | 1 | N | Y/<br>2010-02-19 |
| PPD | 61/<br>F/<br>ASIAN - JAPANESE<br>HERITAGE | LIVER EVENT<br>STOPPING<br>CRITERIA | <b>PPD</b> 68 | 68 | 1 | Υ | Y/<br>2010-04-10 |
| | MEN 2 1110E | LIVER EVENT<br>STOPPING<br>CRITERIA | <b>PPD</b> 134 | 134 | 7 | N | N |

#### **CONFIDENTIAL**

205712

Example :  $PK_F1$  Page 1 of n Protocol : 205712

Population : PK Summary

Figure xx.xx
Box Plot of Plasma Comparative of Geometric Mean (95% CI) with Individual Subjects
CAB Pharmacokinetic Parameters



Programming note: add footnote for treatment A, B.

#### **CONFIDENTIAL**

205712

Example : PK\_F2 Page 1 of n

Protocol : 205712

Population : PK Parameter Summary

Figure xx.xx Geometric Mean Treatment Ratio and 90% CI of CAB Plasma Pharmacokinetic Parameters



Note: The reference lines are at ratios of 0.80, 1.25.

Programming note: add footnote for treatment A, B.